CLINICAL TRIAL: NCT00982228
Title: NN1250-3583: A 52 Week Randomised, Controlled, Open Label, Multicentre, Multinational, Parallel, Treat-to-target Trial Comparing Efficacy and Safety of SIBA and Insulin Glargine Both Administered Once Daily in a Basal-bolus Regimen With Insulin Aspart as Mealtime Insulin in Subjects With Type 1 Diabetes (BEGIN™: BB T1 LONG) / NN1250-3644: An Extension Trial to Trial NN1250-3583 Comparing Safety and Efficacy of NN1250 With Insulin Glargine, Both With Insulin Aspart as Meal-time Insulin, in Type 1 Diabetes (BEGIN™: T1)
Brief Title: Comparison of NN1250 Plus Insulin Aspart With Insulin Glargine Plus Insulin Aspart in Type 1 Diabetes
Acronym: BEGIN™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-3583; 2008-005774-13 (EudraCT Number); U1111-1111-8789 (Other: WHO); 2009-015755-24 (EudraCT Number); U1111-1116-1578 (Other: WHO); NCT01198041 (obsolete NCT alias)
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Results first posted 2015-12-29 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec; Insulin Glargine; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDeg OD (Experimental)
  Interventions: Drug: insulin degludec; Drug: insulin aspart
- IGlar OD (Active Comparator)
  Interventions: Drug: insulin glargine; Drug: insulin aspart

INTERVENTIONS:
Drug: insulin degludec — Injected subcutaneously once daily. Dose was individually adjusted.
  Arms: IDeg OD
Drug: insulin glargine — Injected subcutaneously once daily. Dose individually adjusted.
  Arms: IGlar OD
Drug: insulin aspart — Injected subcutaneously as mealtime insulin. Dose was individually adjusted.

SUMMARY:
This trial is conducted in Africa, Europe and the United States of America (USA).

The aim of the trial is to compare NN1250 (insulin degludec, soluble insulin basal analogue (SIBA)) plus insulin aspart with insulin glargine (IGlar) plus insulin aspart in patients with type 1 diabetes.

The main period is registered internally at Novo Nordisk as NN1250-3583 while the extension period is registered as NN1250-3644.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus for at least 12 months
* Current treatment with any basal bolus insulin for at least 12 months
* HbA1c below or equal to 10.0%
* BMI (Body Mass Index) below or equal to 35.0 kg/m^2
* For the extension trial only: Completion of the 52 week treatment period in trial NN1250-3583 (NCT00982228)

Exclusion Criteria:

* Use of any other antidiabetic drug than insulin within the last 3 months
* Cardiovascular disease within the last 6 months
* Uncontrolled treated/untreated severe hypertension
* Recurrent severe hypoglycemia or hypoglycemic unawareness or hospitalisation for diabetic ketoacidosis during the previous 6 months
* Pregnancy, breast-feeding, the intention of becoming pregnant or not using adequate contraceptive measures according to local requirements
* Cancer and medical history of cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 629 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2010-11-08 (Actual); Study Completion 2010-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (80):
- United States (52):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Huntsville, Alabama
  - Novo Nordisk Investigational Site, Peoria, Arizona
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Greenbrae, California
  - Novo Nordisk Investigational Site, Huntington Beach, California
  - Novo Nordisk Investigational Site, La Mesa, California
  - Novo Nordisk Investigational Site, Los Gatos, California
  - Novo Nordisk Investigational Site, Santa Barbara, California
  - Novo Nordisk Investigational Site, Tustin, California
  - Novo Nordisk Investigational Site, Ventura, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Aurora, Colorado
  - Novo Nordisk Investigational Site, Hollywood, Florida
  - Novo Nordisk Investigational Site, Lake Mary, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Lawrenceville, Georgia
  - Novo Nordisk Investigational Site, Honolulu, Hawaii
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Vincennes, Indiana
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Scarborough, Maine
  - Novo Nordisk Investigational Site, Hyattsville, Maryland
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Brockton, Massachusetts
  - Novo Nordisk Investigational Site, Flint, Michigan
  - Novo Nordisk Investigational Site, Livonia, Michigan
  - Novo Nordisk Investigational Site, Eagan, Minnesota
  - Novo Nordisk Investigational Site, Chesterfield, Missouri
  - Novo Nordisk Investigational Site, Jefferson City, Missouri
  - Novo Nordisk Investigational Site, Saint Charles, Missouri
  - Novo Nordisk Investigational Site, Great Falls, Montana
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Dover, New Hampshire
  - Novo Nordisk Investigational Site, Lawrenceville, New Jersey
  - Novo Nordisk Investigational Site, Flushing, New York
  - Novo Nordisk Investigational Site, Rochester, New York
  - Novo Nordisk Investigational Site, Chapel Hill, North Carolina
  - Novo Nordisk Investigational Site, Raleigh, North Carolina
  - Novo Nordisk Investigational Site, Columbus, Ohio
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Rapid City, South Dakota
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Lubbock, Texas
  - Novo Nordisk Investigational Site, Round Rock, Texas
  - Novo Nordisk Investigational Site, St. George, Utah
  - Novo Nordisk Investigational Site, Renton, Washington
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- France (7):
  - Novo Nordisk Investigational Site, Boisguillaume
  - Novo Nordisk Investigational Site, Brest
  - Novo Nordisk Investigational Site, Grenoble
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Montpellier
  - Novo Nordisk Investigational Site, Nice
  - Novo Nordisk Investigational Site, Paris
- Germany (5):
  - Novo Nordisk Investigational Site, Aschaffenburg
  - Novo Nordisk Investigational Site, Bad Kreuznach
  - Novo Nordisk Investigational Site, Dormagen
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Saint Ingbert
- Russia (6):
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Novosibirsk
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Saint-Peterburg
  - Novo Nordisk Investigational Site, Tyumen
  - Novo Nordisk Investigational Site, Yaroslavl
- South Africa (2):
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Cape Town, Western Cape
- United Kingdom (8):
  - Novo Nordisk Investigational Site, Aberdeen
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, Bradford
  - Novo Nordisk Investigational Site, Glasgow
  - Novo Nordisk Investigational Site, Guildford
  - Novo Nordisk Investigational Site, Leeds
  - Novo Nordisk Investigational Site, Llantrisant
  - Novo Nordisk Investigational Site, Sheffield

REFERENCES:
- [Result] Ratner RE, Gough SC, Mathieu C, Del Prato S, Bode B, Mersebach H, Endahl L, Zinman B. Hypoglycaemia risk with insulin degludec compared with insulin glargine in type 2 and type 1 diabetes: a pre-planned meta-analysis of phase 3 trials. Diabetes Obes Metab. 2013 Feb;15(2):175-84. doi: 10.1111/dom.12032. Epub 2012 Dec 3. PMID 23130654
- [Result] Heller S, Mathieu C, Kapur R, Wolden ML, Zinman B. A meta-analysis of rate ratios for nocturnal confirmed hypoglycaemia with insulin degludec vs. insulin glargine using different definitions for hypoglycaemia. Diabet Med. 2016 Apr;33(4):478-87. doi: 10.1111/dme.13002. Epub 2015 Dec 13. PMID 26484727
- [Result] Sorli C, Warren M, Oyer D, Mersebach H, Johansen T, Gough SC. Elderly patients with diabetes experience a lower rate of nocturnal hypoglycaemia with insulin degludec than with insulin glargine: a meta-analysis of phase IIIa trials. Drugs Aging. 2013 Dec;30(12):1009-18. doi: 10.1007/s40266-013-0128-2. PMID 24170235
- [Result] Einhorn D, Handelsman Y, Bode BW, Endahl LA, Mersebach H, King AB. PATIENTS ACHIEVING GOOD GLYCEMIC CONTROL (HBA1c <7%) EXPERIENCE A LOWER RATE OF HYPOGLYCEMIA WITH INSULIN DEGLUDEC THAN WITH INSULIN GLARGINE: A META-ANALYSIS OF PHASE 3A TRIALS. Endocr Pract. 2015 Aug;21(8):917-26. doi: 10.4158/EP14523.OR. Epub 2015 Jun 29. PMID 26121451
- [Result] Russell-Jones D, Gall MA, Niemeyer M, Diamant M, Del Prato S. Insulin degludec results in lower rates of nocturnal hypoglycaemia and fasting plasma glucose vs. insulin glargine: A meta-analysis of seven clinical trials. Nutr Metab Cardiovasc Dis. 2015 Oct;25(10):898-905. doi: 10.1016/j.numecd.2015.06.005. Epub 2015 Jun 18. PMID 26232910
- [Result] Vora J, Christensen T, Rana A, Bain SC. Insulin degludec versus insulin glargine in type 1 and type 2 diabetes mellitus: a meta-analysis of endpoints in phase 3a trials. Diabetes Ther. 2014 Dec;5(2):435-46. doi: 10.1007/s13300-014-0076-9. Epub 2014 Aug 1. PMID 25081590
- [Result] Aye MM, Atkin SL. Patient safety and minimizing risk with insulin administration - role of insulin degludec. Drug Healthc Patient Saf. 2014 Apr 30;6:55-67. doi: 10.2147/DHPS.S59566. eCollection 2014. PMID 24812526
- [Result] Heller S, Buse J, Fisher M, Garg S, Marre M, Merker L, Renard E, Russell-Jones D, Philotheou A, Francisco AM, Pei H, Bode B; BEGIN Basal-Bolus Type 1 Trial Investigators. Insulin degludec, an ultra-longacting basal insulin, versus insulin glargine in basal-bolus treatment with mealtime insulin aspart in type 1 diabetes (BEGIN Basal-Bolus Type 1): a phase 3, randomised, open-label, treat-to-target non-inferiority trial. Lancet. 2012 Apr 21;379(9825):1489-97. doi: 10.1016/S0140-6736(12)60204-9. PMID 22521071
- [Result] Evans M, Chubb B, Gundgaard J. Cost-effectiveness of Insulin Degludec Versus Insulin Glargine in Adults with Type 1 and Type 2 Diabetes Mellitus. Diabetes Ther. 2017 Apr;8(2):275-291. doi: 10.1007/s13300-017-0236-9. Epub 2017 Feb 16. PMID 28210866
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 79 sites in 6 countries: France (6), Germany (5), Russia (7), South Africa (3), United Kingdom (U.K.) (6) and United States (U.S.) (52).
Pre-assignment Details: All subjects who completed the 52-week main trial (NN1250-3583, NCT00982228) and were found to be eligible for the extension trial were offered to participate in the 52-week extension trial (NN1250-3644).
Groups:
- IDeg OD: Insulin degludec (IDeg) was given subcutaneously (s.c.) once daily (OD) in the evening in combination with insulin aspart (IAsp) as meal time insulin. IDeg was given for 52 weeks in the main period and for an additional 52 weeks in the extension period.
- IGlar OD: Insulin glargine (IGlar) was given s.c. once daily (OD) according to approved labelling in combination with insulin aspart (IAsp) as meal time insulin. IGlar was given for 52 weeks in the main period and for additional 52 weeks in the extension period.
Period: Main: Week 0 to 52 (NN1250-3583)
Arm/Group | IDeg OD | IGlar OD
Started | 472 | 157
Full Analysis Set | 472 | 157
Exposed | 472 | 154 (Three subjects withdrew prior to exposure to trial drug)
Completed | 404 | 137
Not Completed | 68 | 20
Not completed — Adverse Event | 12 | 2
Not completed — Lack of Efficacy | 2 | 0
Not completed — Protocol Violation | 11 | 2
Not completed — Withdrawal criteria | 15 | 3
Not completed — Unclassified | 28 | 13
Period: Extension: Week 53 to 104 (NN1250-3644)
Arm/Group | IDeg OD | IGlar OD
Started | 351 (Fifty-three subjects from the main trial did not continue into the extension) | 118 (Nineteen subjects from the main trial did not continue into the extension)
Completed | 330 | 113
Not Completed | 21 | 5
Not completed — Adverse Event | 3 | 2
Not completed — Lack of Efficacy | 1 | 0
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal criteria | 5 | 0
Not completed — Unclassified | 11 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDeg OD | IGlar OD | Total
Number analyzed (Participants) | 472 | 157 | 629
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (13.7) | 43.7 (13.3) | 43.0 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194 | 67 | 261
  Male | 278 | 90 | 368
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 7.7 (0.9) | 7.7 (1.0) | 7.7 (1.0)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 9.1 (4.0) | 9.7 (4.4) | 9.3 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Main Trial (Primary Endpoint): Change in Glycosylated Haemoglobin (HbA1c) After 52 Weeks of Treatment
Description: Change from baseline in HbA1c after 52 weeks of treatment
Time Frame: Week 0, Week 52
Population: The full analysis set (FAS) included all randomised subjects and missing data was imputed using LOCF (last observation carried forward).
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 472 | 157
percentage of glycosylated haemoglobin | -0.40 (0.73) | -0.39 (0.84)

2. Primary Outcome: Extension Trial (Primary Endpoint): Rate of Treatment Emergent Adverse Events (AEs)
Description: Corresponds to rate of AEs per 100 patient years of exposure. Severity assessed by investigator. Mild: no or transient symptoms, no interference with subject's daily activities. Moderate: marked symptoms, moderate interference with subject's daily activities. Severe: considerable interference with subject's daily activities, unacceptable. Serious AE: AE that at any dose results in any of the following: death, a life-threatening experience, in-subject hospitalization/prolongation of existing hospitalisation, persistent/significant disability/incapacity/congenital anomaly/birth defect.
Time Frame: Week 0 to Week 104 + 7 days follow up
Population: Safety analysis set (SAS) included all subjects who received at least one dose of the investigational product or its comparator in the main trial including subjects carried through to the extension trial.
Measure: Number; unit: Events/100 years of patient exposure
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 472 | 154
Events/100 years of patient exposure
  Adverse events (AE) | 383 | 374
  Serious AE | 14 | 17
  Severe AE | 22 | 26
  Moderate AE | 105 | 106
  Mild AE | 256 | 242
  Fatal AE | 1 | 1

3. Primary Outcome: Extension Trial (Primary Endpoint): Rate of Confirmed Hypoglycaemic Episodes
Description: Rate of confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes are defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes are defined as able to treat her/himself and plasma glucose below 3.1 mmol/L.
Time Frame: Week 0 to Week 104 + 7 days follow up
Population: The SAS included all subjects who received at least one dose of the investigational product or its comparator in the main trial including subjects carried through to the extension trial.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 472 | 154
Episodes/100 years of patient exposure | 3750 | 3743

4. Secondary Outcome: Extension Trial (Primary Endpoint): Rate of Nocturnal Confirmed Hypoglycaemic Episodes
Description: Rate of confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes are defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes are defined as able to treat her/himself and plasma glucose below 3.1 mmol/L. Nocturnal hypoglycaemic episodes are defined as occuring between 00:01 and 05:59 a.m.
Time Frame: Week 0 to Week 104 + 7 days follow up
Population: as for outcome 3
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 472 | 154
Episodes/100 years of patient exposure | 390 | 532

5. Primary Outcome: Extension Trial (Primary Endpoint): Cross-reacting Antibodies to Human Insulin
Description: The unit for measuring antibody levels is amount of tracer bound to the antibodies in the precipitate (B) expressed in percentage of the total amount of tracer (T) added to the mixture (%B/T). Samples were taken before 1st dosing and after a 1-week wash-out period.
Time Frame: Week 0, Week 106
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: %B/T
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 335 | 111
%B/T | 11.3 (15.6) | 11.0 (16.0)

6. Secondary Outcome: Extension Trial (Secondary Endpoint): Change in Glycosylated Haemoglobin (HbA1c) After 104 Weeks of Treatment
Description: Change from baseline in HbA1c after 104 weeks of treatment
Time Frame: Week 0, Week 104
Population: The FAS included all randomised subjects in the main trial including subjects carried through to the extension trial and missing data was imputed using LOCF.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 472 | 157
percentage of glycosylated haemoglobin | -0.27 (0.75) | -0.24 (0.86)

7. Secondary Outcome: Extension Trial (Secondary Endpoint): Mean of 9-point Self Measured Plasma Glucose Profile (SMPG) at Week 104 of Treatment
Description: Mean of 9-point self-measured plasma glucose profile (SMPG) after 104 weeks of treatment. Plasma glucose measured: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after start of dinner, bedtime, at 4 am and before breakfast.
Time Frame: Treatment week 104
Population: The FAS included all randomised subjects in the main trial including subjects carried through to the extension trial and missing data was imputed using LOCF. For 12 subjects all 9-point SMPG values were missing.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 463 | 154
mmol/L | 8.0 (2.2) | 8.1 (2.2)

8. Secondary Outcome: Main Trial (Secondary Endpoint): Rate of Confirmed Hypoglycaemic Episodes
Description: as for outcome 3
Time Frame: Week 0 to Week 52 + 7 days follow up
Population: The SAS included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 472 | 154
Episodes/100 years of patient exposure | 4254 | 4018

9. Secondary Outcome: Main Trial (Secondary Endpoint): Rate of Nocturnal Confirmed Hypoglycaemic Episodes
Description: as for outcome 4
Time Frame: Week 0 to Week 52 + 7 days follow up
Population: The SAS included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 472 | 154
Episodes/100 years of patient exposure | 441 | 586

10. Secondary Outcome: Main Trial (Secondary Endpoint): Mean of 9-point Self Measured Plasma Glucose Profile (SMPG) at Week 52
Description: Mean of 9-point self-measured plasma glucose profile (SMPG) after 52 weeks of treatment. Plasma glucose measured: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after start of dinner, bedtime, at 4 am and before breakfast.
Time Frame: Week 52
Population: The FAS included all randomised subjects and missing data was imputed using LOCF. For 7 subjects all 9-point SMPG values were missing.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDeg OD | IGlar OD
Number analyzed (Participants) | 467 | 155
mmol/L | 8.1 (2.3) | 8.3 (2.4)

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a time frame of 104 weeks + 1 week after last dose in main trial + 1 more week after last dose in extension trial.
Description: The SAS included all subjects who received at least one dose of the investigational product or its comparator.
Arm/Group | IDeg OD | IGlar OD
Serious Adverse Events (participants affected / at risk) | 71/472 | 29/154
Other Adverse Events (participants affected / at risk) | 353/472 | 118/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg OD (N=472) | IGlar OD (N=154)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diabetic gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary gland calculus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pulmonary tuberculoma (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incorrect dose administered (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 27 (38) | 7 (10)
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 15 (20) | 4 (4)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Allergy to animal (Immune system disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Accidental Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon Rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gallbladder cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg OD (N=472) | IGlar OD (N=154)
Diarrhoea (Gastrointestinal disorders) | 39 (44) | 9 (12)
Nausea (Gastrointestinal disorders) | 40 (57) | 14 (18)
Vomiting (Gastrointestinal disorders) | 25 (26) | 11 (15)
Bronchitis (Infections and infestations) | 38 (46) | 11 (17)
Gastroenteritis (Infections and infestations) | 44 (49) | 9 (10)
Influenza (Infections and infestations) | 44 (53) | 17 (19)
Nasopharyngitis (Infections and infestations) | 160 (284) | 51 (105)
Sinusitis (Infections and infestations) | 58 (93) | 23 (31)
Upper respiratory tract infection (Infections and infestations) | 122 (208) | 31 (48)
Urinary tract infection (Infections and infestations) | 35 (40) | 12 (16)
Wrong drug administered (Injury, poisoning and procedural complications) | 31 (35) | 6 (6)
Hypoglycaemia (Metabolism and nutrition disorders) | 44 (70) | 13 (18)
Headache (Nervous system disorders) | 84 (162) | 22 (39)
Cough (Respiratory, thoracic and mediastinal disorders) | 33 (37) | 17 (19)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 34 (46) | 14 (19)
Seasonal allergy (Immune system disorders) | 10 (11) | 10 (10)
Gastrointestinal viral (Infections and infestations) | 25 (27) | 6 (9)
Back Pain (Musculoskeletal and connective tissue disorders) | 33 (46) | 9 (15)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 17 (18) | 11 (13)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 22 (25) | 9 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.